CLINICAL TRIAL: NCT02065258
Title: Comparison Between Breathing and Aerobic Exercises on Clinical Control, Psychosocial Morbidity, Thoracoabdominal Kinematics, and Airway Inflammation in Patients With Moderate-to-severe Asthma: a Randomized Trial
Brief Title: Breathing Versus Aerobic Exercises on Asthma Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Breathing vs. aerobic exercise; 2009538179 (Other Grant/Funding Number: São Paulo Research Foundation)
Record Dates: First submitted 2014-02-03; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: Asthma, Clinical control, Exercise
MeSH Terms: conditions — Asthma; Motor Activity | interventions — Breathing Exercises; Yoga; Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Breathing Exercise (Active Comparator): It will be based on Yoga´s breathing technique (Eliade, 1996) and will be focus on to stimulate nasal and diaphragmatic breathings, to increase expiratory time, to slow respiratory flow and to regulate the breathing rhythm. Breathing exercises will be divided into 3 phases (lasting one month each) with progressive intensity every 8 sessions and will be part of the routine of breathing exercises the following exercises: I) Kapalabhati ; II) Uddhiyana ;III) Surya Bedhana
  Interventions: Other: Breathing exercise
- Aerobic Exercise (Active Comparator): Exercise will be performed on a treadmill, with the initial intensity of 60% of the maximum predicted heart rate for patient´s age (Tanaka et al, 2001) reaching a maximal of 80% during the training. The intensity values will be calculated using Karvonen's formule (1957).Aerobic training sessions that will consist in 40 minutes divided in 5 minutes of warm-up, 35 minutes of aerobic training and 5 minutes of cool down. Exercise intensity will be increased if the patient do not present any increase in asthma symptoms during the exercise for 2 consecutive training days. The program will be performed twice a week, for 3 months.
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Breathing exercise — It will be based on Yoga´s breathing technique (Eliade, 1996) and will be focus on to stimulate nasal and diaphragmatic breathings, to increase expiratory time, to slow respiratory flow and to regulate the breathing rhythm. Breathing exercises will be divided into 3 phases (lasting one month each) with progressive intensity every 8 sessions.
  All participants will be required to maintain their normal medical regimens during the interventions. Will be part of the routine of breathing exercises the following exercises: I) Kapalabhati, II) Uddhiyana
  Other Names: Yoga
  Arms: Breathing Exercise
Other: Aerobic exercise — Exercise will be performed on a treadmill (Imbramed Export Plus, Brazil) with the initial intensity of 60% of the maximum predicted heart rate for patient´s age (Tanaka et al, 2001) reaching a maximal of 80% during the training. The intensity values will be calculated using Karvonen's formule (1957). Exercise intensity will be increased if the patient do not present any increase in asthma symptoms during the exercise for 2 consecutive training days. Before and after every session, patients will perform a peak expiratory flow test and if values were lower than 70% of the patient´s maximum value, they will be advised to use the rescue dose of bronchodilator prescribed the their physician
  Other Names: Aerobic training
  Arms: Aerobic Exercise

SUMMARY:
Background: Asthma is a chronic inflammatory airway disease characterized by reversible obstruction, inflammation and hyperresponsiveness to different stimulus. Aerobic and breathing exercises have been demonstrated to benefit asthmatic patients; however, there is no evidence comparing the effectiveness of the treatments. Objective: To compare the effects of aerobic and breathing exercises on clinical control (primary outcome), psychosocial morbidity and daily life physical activity (secondary outcome) in patients with moderate-to-severe persistent asthma. In addition, thoracoabdominal kinematics, heart rate variability and airway and systemic inflammation will be evaluated. The initial hypothesis will be that both exercises present improved clinical control of asthma. Methods: Forty-eight asthmatic adults will be randomly divided into 2 groups: aerobic (AG) and breathing exercises (BG). All treatments will be performed twice a week for 3 months, totalizing 24 sessions of 40 minutes each. Both groups will complete an educational program consisting of 2 classes at the beginning of the interventions. Before and after interventions, the following parameters will be quantified: clinical control, health related quality of life, levels of anxiety and depression, maximal exercise capacity, autonomic nervous imbalance, daily living physical activity, thoracoabdominal kinematics, inflammatory cells in the sputum, fraction of exhaled nitric oxide (FENO) and systemic inflammatory cytokines. Asthma symptoms will be quantified monthly using diaries. Kolmogorov-Smirnov test will be used to analyze the data normality, and a two-way ANOVA with repeated measures with appropriate post hoc test (Student Newman Keuls) will be used to compare the inter and intra-groups differences

DETAILED DESCRIPTION:
Both groups completed an educational program that consisted of two classes held once a week, each lasting 2 hours. Presentations and group discussions were done, including information about asthma pathophysiology, medication skills, self-monitoring techniques, and environmental control and avoidance strategies.

ELIGIBILITY:
Inclusion Criteria:

* Asthma moderate and severe
* Asthma will diagnosed (Global Initiative for Asthma -GINA)
* Body Mass Index <35 kg/ m2
* Sedentary
* Medical treatment, for at least 6 months
* Clinically stable

Exclusion Criteria:

* Smokers
* Cardiac disease
* Chronic Obstructive Pulmonary Disease
* Active Cancer
* Pregnant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-02 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change from Clinical Control | After 3 months of intervetion
  Clinical control will be evaluated by Asthma Control Questionnaire (ACQ)

SECONDARY OUTCOMES:
Change from psychosocial morbidity | After 3 months of intervetion
  The psychosocial morbidity will be quantified by health factors related to quality of life (Asthma quality of life questionnaire- AQLQ) and depression and anxiety levels (HAD score)
Change from Daily life physical activity (DLPA) | After 3 months of intervetion
  Daily life physical activity will be assessed using an accelerometer (power Walker SW 610, Japan) that records the total daily number of steps and those performed at moderate intensity ( >110 steps per minute)

OTHER OUTCOMES:
Change from Thoracoabdominal kinematics | After 3 months of intervention
  Thoracoabdominal kinematics will be evaluated by using optoelectronic plethysmography (OEP system, BTS, Italy) as previously described Aliverti et al, 2006.
Change from Heart rate variability | After 3 months of interventions
  Heart rate variability will be assessed using heart rate variability (HRV) by a hert rate monitor ( Polar S810i, Finland) previously validated (Gamelin, Berthoin & Bosquet, 2006).
Change from Airway and systemic inflammation | After 3 months of interventions
  Airway inflammation will be quantified using the induced sputum , exhaled fraction of nitric oxide . Systemic inflammation will be evaluated by level of plasmatic inflammatory mediators Th1 ( IL-6, TNF) , Th2 (IL-4, IL-5 and IL-13) and anti-inflammatory ( IL-10 and IL-1ra)

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PT, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Hospital das Clínicas da FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Evaristo KB, Mendes FAR, Saccomani MG, Cukier A, Carvalho-Pinto RM, Rodrigues MR, Santaella DF, Saraiva-Romanholo BM, Martins MA, Carvalho CRF. Effects of Aerobic Training Versus Breathing Exercises on Asthma Control: A Randomized Trial. J Allergy Clin Immunol Pract. 2020 Oct;8(9):2989-2996.e4. doi: 10.1016/j.jaip.2020.06.042. Epub 2020 Aug 6. PMID 32773365
- [Derived] Evaristo KB, Saccomani MG, Martins MA, Cukier A, Stelmach R, Rodrigues MR, Santaella DF, Carvalho CR. Comparison between breathing and aerobic exercise on clinical control in patients with moderate-to-severe asthma: protocol of a randomized trial. BMC Pulm Med. 2014 Oct 17;14:160. doi: 10.1186/1471-2466-14-160. PMID 25326140